CLINICAL TRIAL: NCT06225297
Title: Evaluation of Vector and Chemoprevention-based Interventions to Reduce Malaria Burden in Urban Daaras of Touba, Senegal
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Executive order signed on January 20th 20254 to "reevaluate and realign US foreign aid", resulting in USAID funding freeze
Sponsor: PATH (Other)
Collaborators: L'université de Thiès (Other); University of California, San Francisco (Other); Tulane University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RES-00634
Record Dates: First submitted 2024-01-08; First posted 2024-01-25 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Study participants, community health workers, and study field staff will not be blinded to intervention assignment. However, the trial statistician and laboratory technicians carrying out subsequent analyses in reference laboratories will remain blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention clusters (Experimental): will receive the following interventions:
  1. Distribution of meganets, defined as conventional insecticide-treated nets (ITNs) sewn together to adapt to taalibés sleeping conditions
  2. Three monthly cycles of targeted chemoprevention with dihydroartemisinin-piperaquine (DHA-PQ) for all daara residents, regardless of resident age
  3. Social behavior change (SBC) to promote intervention uptake
  Interventions: Combination Product: Intervention package
- Control clusters (No Intervention): will receive standard-of-care malaria interventions, which include:
  1. Distribution of conventional ITNs
  2. Three monthly cycles of SMC with sulfadoxine-pyrimethamine- amodiaquine (SP-AQ) given to children 3-120 months

INTERVENTIONS:
Combination Product: Intervention package — Intervention package will include vector control through meganets (multiple insecticide-treated mosquito nets sewn together), seasonal malaria chemoprevention (SMC) extended to all ages using DHA-PQ, and behavior change communication.
  Arms: Intervention clusters

SUMMARY:
This study aims to evaluate the effectiveness of the use of adapted insecticide-treated mosquito nets combined with extended DHA-PQ-based seasonal chemoprevention for all ages and behavior change communication in reducing the burden of malaria in relation to standards of protection and care among students (taalibés) in the daaras (Koranic schools) of Touba, Senegal.

DETAILED DESCRIPTION:
In Senegal, young children (mostly boys) may be sent to religious schools (daaras) to learn about the Koran and moral and cultural values. The students (talibés) often live and sleep in crowded conditions and as a result, insecticide-treated net (ITN) use is consistently low due to challenges faced in hanging ITNs as well as difficulty covering multiple children sleeping together. This study will consist of a two-arm cluster-randomized controlled trial to evaluate the effectiveness of an intervention package in urban daaras in Touba City, Diourbel region, Senegal.

The intervention package will include vector control through meganets (multiple insecticide-treated mosquito nets sewn together and adapted based on the needs and sleeping situation of the daara), seasonal malaria chemoprevention (SMC) extended to all ages using DHA-PQ, and behavior change communication.

Prior to evaluating an intervention, there will be 1) a mapping of the daaras in Touba City, Diourbel Region of Senegal to observe the various structures and types of daaras in order to select typical daaras for the entomological component, and to inform randomization, 2) human behavior observation (HBO) of students (talibes) and teachers (marabouts) in 2-3 daaras selected through the mapping to help tailor the intervention package, and 3) analysis of mosquito behavior observed through human landing catches.

Two cross-sectional surveys will be conducted, before and after the intervention, which will include an electronic questionnaire to be sent to the taalibés themselves or to their guardians, a temperature reading, an RDT for participants with a fever at the time of the survey, and a fingertip blood sample to assess parasite prevalence (microscopy and PCR). Qualitative surveys will be carried out using a mixed-method design, consisting of a literature review, in-depth individual interviews, focus groups, and on-site observations. Meganet monitoring surveys will be carried out after meganet distribution to assess the attrition and physical integrity of the nets.

Malaria incidence will be determined from records of community health workers assigned to the daaras who have been trained by the Ministry of Health to identify febrile students, test them for malaria using a rapid diagnostic test and treat confirmed cases with an antimalarial medicine. Additional data on students who seek care from health centers in their neighborhood will supplement the data obtained from community health workers.

ELIGIBILITY:
Inclusion criteria for daara:

* Located within the catchment area of Touba Health District
* Located within the catchment area of a health facility with an annual malaria incidence of ≥ 25 cases per 1000 population
* Daara is registered in the health system and the Serigne daara (i.e., daara leader) can provide caregiver consent for taalibé.
* Taalibé population between 29 to 120
* PECAdaara model has been integrated and fully operational
* Willingness of daara leader to participate in the study

Inclusion criteria for receiving DHA-PQ:

* Age ≥ 3 months
* Taalibé of study daara
* Willingness to comply with study procedures
* Provision of informed consent/assent

Additional inclusion criteria for receiving meganets:

- Sleeping in a superimposed area with ≥ 2 people

Exclusion Criteria for receiving DHA-PQ:

* Age < 3 months
* Refusal of informed consent
* Concomitant or recent use of antimalarials within the past two weeks
* Known allergy or hypersensitivity to DHA-PQ
* Confirmed diagnosis of clinical malaria
* Currently taking anti-worm or anti-infection drugs, including cotrimoxazole (BACTRIM), mebendazole, quinolones, sulfonamides (FANSIDAR, MALOXINE), dapsone, colchicine
* Currently taking medications that influence cardiac function or prolong the QTc interval
* Serious or chronic illness, including known HIV infection, heart disease, or severe malnutrition (weight-for-age or mid-upper arm circumference (MUAC) < 3 SD)
* Pregnancy (assessed by history or urine pregnancy test)

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4600 (Estimated)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Difference in cumulative incidence of clinical malaria confirmed by rapid diagnostic test (RDT) between arms | monthly basis over 12 months
  Cumulative incidence will be defined as the number of RDT-confirmed malaria cases per 1000 population in each daara. Cases will be identified from both PECAdaara and health facility registries
Difference in change in prevalence of microscopy-confirmed infection between arms | 12 months
  Prevalence will be defined as the proportion of individuals with microscopy-confirmed infection assessed during the endline survey
Difference in pre-post change in prevalence of PCR-confirmed infection between arms | 12 months
  Prevalence will be defined as the proportion of individuals with PCR-confirmed infection, assessed during cross-sectional surveys

SECONDARY OUTCOMES:
Difference in cumulative incidence of grade 3+ adverse events after drug administration between arms | 12 months
  Defined as the number of grade 3+ AEs divided by the participant population who received at least one dose of drug.
Difference in the cumulative incidence of serious adverse events (SAE) after SMC administration between arms | 12 months
  Adverse events will be classified as serious or non-serious based on standardized AE grading scale
Difference in human behavior on net use before and after ITN/meganet distribution | 12 months
  ITN use (e.g., sleeping under net in the previous night, sleeping indoors versus outdoors) will be assessed during cross-sectional surveys
Difference in indoor and outdoor adjusted human biting rates between arms | 12 months
  The human landing rate will be used as a proxy for the human biting rate (HBR). The HBR data will be integrated with the human behavior observation (HBO) data on net use and sleep patterns data by calculating the hourly adjusted HBR.
Difference in Anopheles biting trends between arms | 12 months
  Anopheles biting trends will be examined by measuring the Anopheles biting times (including peak biting time), biting locations (indoors and outdoors), and vector density (defined as mean number of bites received by one person in one night) during human landing catches
Acceptability of intervention package | 12 months
  Perceptions of intervention package and reasons for participation assessed through qualitative studies conducted throughout the study period
Difference in proportion of refusals between arms | 12 months
  Refusals will be defined as the number of those who refused a specific intervention divided by the number of participants who were targeted and eligible to receive the specific intervention (i.e., chemoprevention and meganets).
Difference in distribution coverage of chemoprevention strategies between arms | 12 months
  Distribution coverage will be defined as the number of persons who received intervention divided by number of those targeted and eligible
Difference in crude coverage of chemoprevention strategies between arms | 12 months
  Crude coverage will be defined using WHO criteria as number of persons who received the intervention divided by number of those who were targeted (regardless of eligibility)
Cost per malaria case averted | 12 months
  Total intervention costs will be calculated in both arms and compared with efficacy measures of malaria incidence to generate the incremental cost effectiveness ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis Ndiaye, Principal Investigator — L'université de Thiès
Locations (1):
- Daaras in Touba, Touba, Senegal

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/97/NCT06225297/ICF_000.pdf